CLINICAL TRIAL: NCT06757439
Title: Effect of Frailty on Spinal Anesthesia-induced Hypotension in Geriatric Patients
Brief Title: Frailty and Spinal Anesthesia-Induced Hypotension in Elderly
Status: Not yet recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Mehmet SARGIN, Associate Professor, Selcuk University
Other Study IDs: 2024-12-1
Record Dates: First submitted 2024-12-19; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Frailty; Spinal Anesthesia
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Frail: CFS Level ≥4
- Non-frail: CFS Level ≤3

SUMMARY:
60 patients aged 65 and older with ASA I-III physical status undergoing elective surgery under spinal anesthesia will be included in the study.

Patients with cardiac arrhythmia, severe heart failure, cerebrovascular disease, or contraindications to neuraxial anesthesia will be excluded. Frailty assessments will be performed using the Clinical Frailty Scale (CFS) version 2.0 by anesthesiologists in preoperative clinics or wards. Participants will be categorized into frail (CFS Level ≥4, Group I) and non-frail (CFS Level ≤3, Group II) groups.

Prior to spinal anesthesia, 8 mL/kg of crystalloids will be administered. Baseline preoperative mean arterial blood pressure (MABP) and heart rate (HR) will be recorded as the average of three measurements in the supine position.

During the study, MABP and HR will be monitored every 2 minutes for the first 20 minutes post-spinal anesthesia, then every 5 minutes until surgery ends. Hypotension (MABP <80% of baseline) will be treated with 5 mg intravenous ephedrine, while bradycardia (HR <50 beats/min) will be treated with 0.5 mg intravenous atropine.

ELIGIBILITY:
Inclusion Criteria:

* 65 and older
* ASA I-III physical status
* Undergoing elective surgery under spinal anesthesia

Exclusion Criteria:

* Patients with cardiac arrhythmia
* Patients with severe heart failure
* Patients with cerebrovascular disease
* Contraindications to neuraxial anesthesia

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Male and female patients aged 65 and over
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-01-20 (Estimated); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Rate of Hypotension | Preoperative baseline, every 2 minutes for the first 20 minutes, and then at 5-minute intervals until the completion of the surgery.
  Hypotension, defined as MABP below 80% of baseline values

SECONDARY OUTCOMES:
Rate of Bradycardia | Preoperative baseline, every 2 minutes for the first 20 minutes, and then at 5-minute intervals until the completion of the surgery.
  Bradycardia defined as HR <50 beats/min
Ephedrine usage | During the procedure
  Necessary use of ephedrine (mg) for patients who develop hypotension
Rate of Nausea and vomiting | up to 24 hours
  Nausea and vomiting Visual analogue scale

IPD SHARING:
Plan to Share IPD: Undecided